CLINICAL TRIAL: NCT01475305
Title: A Phase 1 Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of MEDI-557 in Healthy Adults Intranasally Challenged With Respiratory Syncytial Virus (RSV)
Brief Title: Intranasal Challenge of Healthy Adults With Respiratory Syncytial Virus (RSV)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated as it was determined to not be feasible to complete enrollment and the study within the required timeline and budget.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CD-ID-MEDI-557-1090
Record Dates: First submitted 2011-10-14; First posted 2011-11-21 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: RSV Infection
Keywords: Respiratory Syncytial Virus (RSV); Healthy adults; MEDI-557; Intranasal challenge; Human model
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received single intravenous (IV) dose of placebo matched to MEDI-557 on Day 1 and were inoculated with respiratory syncytial virus (RSV-A) (Memphis-37 strain) as intranasal drops on Day 3.
  Interventions: Drug: Placebo
- MEDI-557 (Experimental): Participants received single IV dose of 30 milligram per kilogram (mg/kg) MEDI-557 on Day 1 and were inoculated with RSV-A (Memphis-37 strain) as intranasal drops on Day 3.
  Interventions: Drug: MEDI-557

INTERVENTIONS:
Drug: Placebo — Participants received single intravenous (IV) dose of placebo matched to MEDI-557 on Day 1 and were inoculated with respiratory syncytial virus (RSV-A) (Memphis-37 strain) as intranasal drops on Day 3.
  Arms: Placebo
Drug: MEDI-557 — Participants received single IV dose of 30 milligram per kilogram (mg/kg) MEDI-557 on Day 1 and were inoculated with RSV-A (Memphis-37 strain) as intranasal drops on Day 3.
  Arms: MEDI-557

SUMMARY:
The primary objective is to evaluate the suitability of the challenge model in measuring the efficacy of MEDI-557 compared to placebo in healthy adult participants for the reduction in the incidence of RSV through 12 days post-RSV challenge with the RSV Memphis-37 strain.

DETAILED DESCRIPTION:
This is designed to be a double-blind, placebo-controlled, randomized study. Approximately 30 participants will be randomized, dosed and followed. Participants will be randomly assigned to receive a single intravenous (IV) dose of MEDI-557 or placebo. Participants will be inoculated with RSV-A. Participants will be followed for efficacy for 12 days post-RSV challenge. Safety follow-up will be approximately 12 months from randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by medical history and physical examination.
2. Age 19 through 38 years at the time of screening.
3. Written informed consent and any locally required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
4. Weight less than or equal to (<=) 10 kilogram (kg) with body mass index (BMI) less than (<) 32 kilogram per meter square (kg/m^2).
5. Normotensive (systolic blood pressure [BP] <150 millimeters of mercury (mmHg) and diastolic BP < 90 mmHg).
6. Females of childbearing age using contraception.
7. Males who are sexually active with a female partner of childbearing potential, using contraception.
8. Sero-suitable (that is, low serum RSV neutralizing antibody titre) for RSV infection.

Exclusion Criteria:

Current medical conditions as follows:

1. Clinical evidence of chronic pulmonary disease or any use of a bronchodilator or other asthma medication.
2. Current smoker unwilling/unable to desist for the quarantine phase of the study.
3. History or clinical evidence of recurrent lower respiratory tract infection.
4. Evidence of infection with hepatitis A, B, or C virus or human immunodeficiency virus (HIV) by serology.

   Medical history as follows:
5. History of immunodeficiency.
6. History of chronic sinusitis.
7. History of frequent epistaxis.
8. History of or current diagnosis of diabetes.
9. Prior/concomitant therapy including

   * Receipt of any systemic chemotherapeutic agent at any time;
   * Receipt of systemic glucocorticoids within 1 month, or any other immunosuppressive drug within 6 months prior to challenge.
   * Receipt of any investigational drug within 6 months prior to dose or concurrent enrolment in another clinical study.
   * Prior participation in a clinical trial of any experimental RSV viral challenge delivered directly to the respiratory tract at any time, or any other respiratory virus challenge within 1 year prior to dose.
10. Nursing mother.
11. Alcohol or drug addiction/abuse within the past 2 years.
12. A positive urine Class A drug or alcohol screen unless there is a medical reason.
13. History of seasonal hay fever or seasonal allergies.
14. Employees of the clinical study site or sponsor, any other individuals involved with the conduct of the study, or immediate family members of such individuals.
15. Health care workers anticipated to have patient contact within 2 weeks after viral challenge.
16. Participants who, for an additional 2 weeks after discharge from the isolation facility, are likely to have contact with a household member or close contact with someone who is: (a) less than 3 years of age; (b) any person with any known immunodeficiency; (c) any person receiving immunosuppressant medications; (d) any person undergoing or soon to undergo cancer chemotherapy within 28 days of challenge; (e) any person who has diagnosed emphysema or COPD, is elderly residing in a nursing home, or with severe lung disease or medical condition; or (f) any person who has received a transplant (bone marrow or solid organ).
17. As a result of the medical interview, physical examination, or screening investigations, the investigator(s) considers the participant unfit for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10-20 (Actual); Primary Completion 2011-12-03 (Actual); Study Completion 2012-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Jafri, MD, Study Director — MedImmune LLC
Locations (1):
- Research Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 90 participants were screened, out of these, 7 participants were randomized and completed the study.
Period: Overall Study
Arm/Group | Placebo | MEDI-557
Started | 4 | 3
End of Quarantine, Day 15 | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI-557 | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.5 (4.4) | 28.0 (9.5) | 26.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Developing Respiratory Syncytial Virus (RSV) Infection Post-RSV Challenge Measured by Plaque Assay Culture
Description: RSV infection is defined as positive plaque assay culture sample for greater than or equal to (>=) 1 day through 12 days post-RSV challenge. A sample was determined positive if log10 plaque-forming units per milliliter [pfu/mL] greater than or equal lower limit of quantitation (LLOQ; 1.69 log10 pfu/mL) and 2 of the 3 replicates must have greater than (>) 0 pfu/mL.
Time Frame: From Day 4 to Day 15
Population: Population for RSV Incidence included all participants who received both the investigational product and RSV challenge.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 3 | 3
percentage of participants | 66.7 | 0.0
Statistical Analysis 1: Comparison: Placebo vs MEDI-557; Test type: Superiority or Other; Relative Risk = 0.00, 95% CI 2-sided [0.00 to 2.05] — Relative risk was calculated as the proportion of participants with RSV infection in the MEDI-557 arm divided by the proportion of participants with RSV infection in the placebo arm

2. Secondary Outcome: Percentage of Participants Developing Respiratory Syncytial Virus (RSV) Infection Post-RSV Challenge Measured by Quantitative Real-Time Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), Direct Fluorescent Antibody (DFA), And by Any Method
Description: RSV infection defined as positive quantitative real-time RT-PCR (RSV-A only) sample for >= 2 consecutive days through 12 days post-RSV challenge. A sample was determined positive if log10 copies/ml >= limit of quantitation (LLOQ; 2.80 log10 copies/mL). RSV infection defined as positive DFA sample for >= 2 consecutive days through 12 days post-RSV challenge. RSV infection by any method included positive plaque assay culture sample for >=1 day through 12 days post-RSV challenge, or positive quantitative real-time RT-PCR (RSV-A only) sample for >= 2 consecutive days through 12 days post-RSV challenge, or positive DFA sample for >=2 consecutive days through 12 days post-RSV challenge.
Time Frame: From Day 4 to Day 15
Population: Population for RSV Incidence included all participants who received both the investigational product and RSV challenge.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 3 | 3
percentage of participants
  RSV infection by quantitative real-time RT-PCR | 66.7 | 66.7
  RSV infection by DFA | 66.7 | 0.0
  RSV infection by Any Method | 66.7 | 66.7
Statistical Analysis 1: Comparison: Placebo vs MEDI-557; RSV infection by quantitative real-time RT-PCR; Test type: Superiority or Other; Relative Risk = 1.00, 95% CI 2-sided [0.16 to 6.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs MEDI-557; RSV infection by DFA; Test type: Superiority or Other; Relative Risk = 0.00, 95% CI 2-sided [0.00 to 2.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs MEDI-557; RSV infection by Any Method; Test type: Superiority or Other; Relative Risk = 1.00, 95% CI 2-sided [0.16 to 6.24] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Viral Load AUC0-t by Plaque Assay Culture
Description: RSV infection by plaque assay culture defined as positive sample for >= 1 day through 12 days post-RSV challenge.
Time Frame: From Day 5 through Day 31
Population: Population for RSV Plaque Assay Culture Virology included all participants who received both investigational product and RSV challenge and were positive for RSV by plaque assay culture (defined as positive sample for >=1 day through 12 days post-RSV challenge).
Measure: Mean (Standard Deviation); unit: log10 pfu*day/mL
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 2 | 0
log10 pfu*day/mL | 42.165 (3.305) |

4. Secondary Outcome: Mean Viral Load AUC0-t by Realtime Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
Description: RSV infection by plaque assay culture defined as positive sample for >= 2 consecutive days through 12 days post-RSV challenge.
Time Frame: From Day 5 through Day 31
Population: Population for RSV Quantitative Real-Time RT-PCR Virology included all participants who received both the investigational product and RSV challenge and were positive for RSV-A by quantitative real-time RT-PCR (defined as positive samples for >= 2 consecutive days through 12 days post-RSV challenge).
Measure: Mean (Standard Deviation); unit: log10 copies*day/mL
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 2 | 2
log10 copies*day/mL | 100.04 (7.000) | 65.708 (1.488)

5. Secondary Outcome: Mean Nasal RSV Peak as Measured by Plaque Assay Culture
Description: RSV infection by plaque assay culture defined as positive sample for >= 1 day through 12 days post-RSV challenge. log10 pfu/mL = log10 plaque-forming unit per milliliter.
Time Frame: From Day 5 through Day 31
Population: Population for RSV Plaque Assay Culture Virology included all participants who received both investigational product and RSV challenge and were positive for RSV by plaque assay culture (defined as positive sample for >= 1 day through 12 days post-RSV challenge).
Measure: Mean (Standard Deviation); unit: log10 pfu/mL
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 2 | 0
log10 pfu/mL | 4.150 (0.521) |

6. Secondary Outcome: Mean Nasal RSV Peak as Measured by Quantitative Realtime Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
Description: as for outcome 4
Time Frame: From Day 5 through Day 31
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 2 | 2
log10 copies/mL | 7.700 (0.453) | 4.260 (0.863)

7. Secondary Outcome: Duration of Respiratory Syncytial Virus (RSV) Viral Shedding
Description: Duration of viral shedding defined as the number of days from the first sample positive by any assay (that is, plaque assay culture, quantitative real-time (RT-PCR), or direct fluorescent Antibody (DFA) to the last sample positive by any assay.
Time Frame: From Day 5 through Day 31
Population: Population for RSV Incidence by any Viral Assay included all participants who received both the investigational product and RSV challenge and were positive for RSV by plaque assay culture, quantitative real-time RT-PCR, or DFA.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 2 | 2
days | 10.0 (0.0) [10 to 10] | 6.5 (4.5) [2 to 11]

8. Secondary Outcome: Mean Serum MEDI-557 Concentration Through Day 360
Description: MEDI-557 serum concentrations were summarized by each sampling point [LLOQ for MEDI-557 concentration assay was 1.56 microgram per millilitre (μg/mL) for serum].
Time Frame: Pre-dose (Day 1); 1,4 and 8 hours post-dose on Day 1 and post-dose on Days 2, 3, 5, 7, 9, 11, 15, 31, 61, 91, 120, 150, 180, 240, 300 and 360
Population: Population for PK included all participants who received a full dose of investigational product and had >= 1 post-baseline measurement for PK. Here n = participants evaluable for specified categories, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (ug/mL)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
microgram per milliliter (ug/mL)
  Day 1 (pre-dose) (n=3) | 0.000 (0.000)
  1 hr Post-dose (n=3) | 498.730 (6.615)
  4 hr Post-dose (n=3) | 462.937 (40.212)
  8 hr Post-dose (n=3) | 458.413 (40.613)
  Day 2 (n=3) | 407.627 (13.420)
  Day 3 (n=3) | 343.283 (48.078)
  Day 5 (n=3) | 298.020 (48.966)
  Day 7 (n=3) | 287.917 (39.276)
  Day 9 (n=3) | 293.897 (33.128)
  Day 11(n=3) | 265.107 (24.076)
  Day 15 (n=3) | 252.327 (16.091)
  Day 31 (n=3) | 252.177 (23.225)
  Day 61 (n=2) | 180.505 (6.442)
  Day 91 (n=3) | 131.053 (4.571)
  Day 120 (n=3) | 106.040 (10.023)
  Day 150 (n=3) | 75.583 (11.258)
  Day 180 (n=3) | 65.443 (5.897)
  Day 240 (n=2) | 43.875 (6.428)
  Day 300 (n=3) | 31.353 (5.731)
  Day 360 (n=3) | 20.343 (4.138)

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of MEDI-557
Description: The Cmax is the maximum observed serum concentration of MEDI-557.
Time Frame: as for outcome 8
Population: Population for PK included all participants who received a full dose of investigational product and had >= 1 post-baseline measurement for PK.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/ml)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
microgram per milliliter (mcg/ml) | 504.0433 (6.6189)

10. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of MEDI-557
Description: The Tmax is defined as actual sampling time to reach maximum observed MEDI-557 concentration.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
Day | 0.162 (0.068)

11. Secondary Outcome: Serum Half Life (t1/2) of MEDI-557
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
Day | 94.0029426 (93.8412056)

12. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of MEDI-557
Description: The AUC(0-t) is the area under the serum concentration-time curve from time zero to any time 't'.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*microgram per milliliter (d*mcg/ml)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
day*microgram per milliliter (d*mcg/ml) | 34484.8642 (1114.4471)

13. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of MEDI-557
Description: The AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: d*mcg/ml
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
d*mcg/ml | 37266.5740 (1764.7070)

14. Secondary Outcome: Volume of Distribution at Steady-State (Vss) of MEDI-557
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the serum concentration-time curve from time zero to infinite time.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliliter (ml)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
milliliter (ml) | 6644.3433 (606.4269)

15. Secondary Outcome: Mean Clearance of MEDI-557
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the serum Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]).
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliliter per day (ml/d)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
milliliter per day (ml/d) | 50.3831 (4.6158)

16. Secondary Outcome: Mean Nasal Wash Concentration of MEDI-557 at Respective Time-Points
Description: MEDI-557 nasal wash concentrations were summarized by each sampling point [LLOQ for MEDI-557 concentration assay was 20.00 nanogram per millilitre (ng/mL) for nasal wash].
Time Frame: Pre-dose (Day 1) and post-dose on Days 2, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, and 31
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
nanogram per milliliter (ng/mL)
  Day 1 (pre-dose) | 0.000 (0.000)
  Day 2 | 166.613 (8.257)
  Day 5 | 192.827 (160.257)
  Day 6 | 189.767 (87.745)
  Day 7 | 227.980 (189.806)
  Day 8 | 308.153 (173.823)
  Day 9 | 201.647 (105.288)
  Day 10 | 132.407 (134.702)
  Day 11 | 220.953 (58.505)
  Day 12 | 262.800 (310.692)
  Day 13 | 89.867 (72.249)
  Day 14 | 184.747 (260.718)
  Day 15 | 243.567 (251.884)
  Day 31 | 62.707 (62.348)

17. Secondary Outcome: Maximum Nasal Wash Concentration (Cmax) of MEDI-557
Description: The Cmax is the maximum observed nasal wash concentration of MEDI-557.
Time Frame: Pre-dose (Day 1) and post-dose on Days 2, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, and 31
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
nanogram per milliliter (ng/ml) | 377.9800 (212.2542)

18. Secondary Outcome: Time to Reach Maximum Nasal Wash Concentration (Tmax) of MEDI-557
Description: The Tmax is defined as actual sampling time to reach maximum observed MEDI-557 concentration.
Time Frame: Pre-dose (Day 1) and post-dose on Days 2, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, and 31
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
Day | 9.051 (2.113)

19. Secondary Outcome: Area Under the Nasal Wash Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of MEDI-557
Description: The AUC(0-t) is the area under the nasal wash concentration-time curve from time zero to any time 't'.
Time Frame: Pre-dose (Day 1) and post-dose on Days 2, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, and 31
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*nanogram per milliliter (d*ng/ml)
Arm/Group | MEDI-557
Number analyzed (Participants) | 3
day*nanogram per milliliter (d*ng/ml) | 4541.3636 (3905.7874)

20. Secondary Outcome: Percentage of Participants With Positive Anti-MEDI-557 Antibodies
Description: Anti-drug antibodies in the participants blood sample were detected using a validated immunoassay. Antidrug antibodies to MEDI-557 were defined as a detectable antibody titer with a dilution value of 1:30 or greater.
Time Frame: Day 1 (pre-dose); Day 31, 91, 150, 180, 240, 300 and 360 post-dose
Population: Population for ADA included all participants who received any amount of investigational product and had >= 1 post-baseline measurement for ADA. Here, "n" is number of participants analysed at specific time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 4 | 3
percentage of participants
  Day 1 (pre-dose) (n=4,3) | 0 | 0
  Day 31 (n=4,3) | 0 | 0
  Day 91 (n=4,3) | 0 | 0
  Day 150 (n=3,3) | 0 | 33.3
  Day 180 (n=4,3) | 0 | 66.7
  Day 240 (n=3,2) | 0 | 50.0
  Day 300 (n=4,3) | 0 | 33.3
  Day 360 (n=4,3) | 0 | 0

21. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and Day 360 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Day 1 (immediately following administration of study drug) to Day 360
Population: Safety Population included all participants who received any amount of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 4 | 3
participants
  TEAEs | 1 | 0
  TESAEs | 4 | 3

22. Secondary Outcome: Number of Participants With Vital Signs Abnormalities Reported as Adverse Events (AEs)
Description: Vital signs included temperature, respiration rate, heart rate, blood pressure. Abnormal vital sign parameters included Cardiac Disorders (Bradycardia), Respiratory, Thoracic and Mediastinal Disorders (Tachypnoea, Hyperventilation, Hypopnoea). Participants with abnormalities in these vital Signs investigations recorded as AEs were reported.
Time Frame: From Day 1 through Day 31
Population: Safety Population included all participants who received any amount of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 4 | 3
participants | 3 | 3

23. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Investigations Reported as Adverse Events (AEs)
Description: Laboratory investigations included hematology, coagulation, serum chemistry and urinalysis parameters. Participants with abnormalities in these laboratory investigations recorded as AEs were reported.
Time Frame: From Day 1 through Day 91
Population: Safety Population included all participants who received any amount of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 4 | 3
participants
  Hematology | 0 | 0
  Coagulation | 0 | 0
  Serum chemistry | 0 | 2
  Urinalysis | 0 | 2
  Cardiac enzymes | 1 | 0

24. Secondary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Spirometry Values
Description: Spirometry is a standardized assessment to evaluate lung function. Baseline values for spirometry is defined as the last measure prior to viral challenge. Spirometry assessments included percent predicted forced expiratory volume in 1 second (FEV1), FEV1/forced vital capacity (FVC), and forced expiratory flow (FEF) 25%-75% values.
Time Frame: Days 1, 2, 3 (Baseline), 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 31
Population: Safety Population included all participants who received any amount of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI-557
Number analyzed (Participants) | 4 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day -2 to Day 360
Description: Safety population included all participants who received any amount of investigational product.
Arm/Group | Placebo | MEDI-557
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | MEDI-557 (N=3)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | MEDI-557 (N=3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 2 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (6)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated before an adequate number of subjects were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.